CLINICAL TRIAL: NCT04689022
Title: Predictors of Treatment Failure Among Patients With Gunshot Wounds and Post-traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vasyl' Horoshko (Other)
Collaborators: Bogomolets National Medical University (Other)
Responsible Party: Sponsor-Investigator, Vasyl' Horoshko, Principal Investigator, Bogomolets National Medical University
Organization: Bogomolets National Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BogomoletsNMU
Record Dates: First submitted 2020-12-17; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Gunshot Entry Wound
Keywords: Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Pain Measurement

STUDY DESIGN:
Intervention Model Description: A total of 218 patients completed the study. The Mississippi Scale for Combat-Related PTSD (M-PTSD) was used for assessment of the treatment outcome rate. The risk relation between treatment failure and factors was assessed by a univariate or multivariate logistic regression method, with the model accuracy measured by the AUC - Area under the ROC curve. The odds ratio (OR) was considered for the qualitative factor assessment.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group І received general anesthesia (n=53) (Other): The sedation with constant rate infusion of 1% propofol, 1-4mg/kg/h, guided by Bispectral analysis (60-70 - for regional anesthesia and 40-60 - for the general one). 0.005% fentanyl analgesia was injected, 3-10 mkg/kg or 0.05-0.2 mkg/kg/min during induction; and 2-10 mkg/kg/h for maintaining analgesia, by periodic bolus injection 25-100 mkg or by permanent infusion.
  The postoperative pain management of the I group patients was provided according to the local clinical protocol: paracetamol+/-non-steroid anti-inflammatory drugs +/-opioids.
  The PTSD progress and treatment effectiveness were estimated using the Mississippi Scale for Combat-Related PTSD, anesthesia risks - the American Society of Anesthesiologists classification, pain intensity - the visual analogue scale, neuropathic pain component - the Douleur Neuropathique 4 questions.
  Interventions: Behavioral: Mississippi Scale for Combat-Related PTSD (M-PTSD); Diagnostic Test: visual analogue scale (VAS); Diagnostic Test: Douleur Neuropathique 4 questions (DN4)
- Group II received regional anesthesia: peripheral block was performed (n=73) (Other): The regional anesthesia was guided by ultrasound (apparatus Mindray DP-30 with linear array probe 5-10 MHz). A needle was inserted near the nerve roots and 20-30 ml of 0.5% bupivacaine was injected.
  The postoperative pain management - repeated peripheral block or prolonged regional anesthesia with 0.25% bupivacaine solution.
  The PTSD progress and treatment effectiveness were estimated using the Mississippi Scale for Combat-Related PTSD, anesthesia risks - the American Society of Anesthesiologists classification, pain intensity - the visual analogue scale, neuropathic pain component - the Douleur Neuropathique 4 questions.
  Interventions: Behavioral: Mississippi Scale for Combat-Related PTSD (M-PTSD); Diagnostic Test: visual analogue scale (VAS); Diagnostic Test: Douleur Neuropathique 4 questions (DN4)
- Group III received regional anesthesia with sedation (n=92) (Other): The regional anesthesia was guided by ultrasound (apparatus Mindray DP-30 with linear array probe 5-10 MHz). A needle was inserted near the nerve roots and 20-30 ml of 0.5% bupivacaine was injected.
  The postoperative pain management - repeated peripheral block or prolonged regional anesthesia with 0.25% bupivacaine solution.
  The PTSD progress and treatment effectiveness were estimated using the Mississippi Scale for Combat-Related PTSD, anesthesia risks - the American Society of Anesthesiologists classification, pain intensity - the visual analogue scale, neuropathic pain component - the Douleur Neuropathique 4 questions.
  Interventions: Behavioral: Mississippi Scale for Combat-Related PTSD (M-PTSD); Diagnostic Test: visual analogue scale (VAS); Diagnostic Test: Douleur Neuropathique 4 questions (DN4)

INTERVENTIONS:
Behavioral: Mississippi Scale for Combat-Related PTSD (M-PTSD) — The treatment outcome rate was assessed by the Mississippi Scale for Combat-Related PTSD (M-PTSD). A positive outcome rate is represented with the patient post-discharge positive coping, which corresponds to 94-58 points, observed in 39 patients (17.9%). A treatment failure is regarded as the absent PTSD treatment effect after discharge, which corresponds to 148-113 points, observed in 5 patients (2.3%) and psychic disorders, which correspond to 112-95 points, observed in 174 patients (79,8%).
  Other Names: The PTSD progress and treatment effectiveness were estimated using the Mississippi Scale for Combat-Related PTSD (M-PTSD)
Diagnostic Test: visual analogue scale (VAS) — pain intensity
  Other Names: VAS
Diagnostic Test: Douleur Neuropathique 4 questions (DN4) — neuropathic pain component
  Other Names: DN4

SUMMARY:
The 82.1% treatment failure of post-traumatic stress disorder(PTSD), associated with gunshot wounds, is related to high incidence of chronic pain syndrome as well as resistance to the PTSD treatment. Defining treatment failure predictors among the PTSD patients with gunshot extremity wounds and the following therapy would improve treatment outcomes.

DETAILED DESCRIPTION:
It has been noted that the PTSD in military combatants results from their direct participation in military actions. The study revealed that if a military combatant was wounded during the action operation, his emotional and subjective feelings will 100% lead to the PTSD. Other scientists state about the PTSD remote treatment failure in 80% of the military combatants. The study evidences about 82.1% of the PTSD m-related wounds treatment failure, which was essential for the subsequent studies. Some authors state about treatment effectiveness of psychopharmacological drugs and psychotherapy, which is rather questionable. Traumas and somatic diseases in the PTSD patients are known to accumulate their negative effects. So, definition of the PTSD treatment failure predictors may improve treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* gunshot wounds
* post-traumatic stress disorder
* patients who need anesthesia

Exclusion Criteria:

* the patient has no post-traumatic stress disorder
* the patient has no gunshot wounds

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 218 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Mississippi Scale for Combat-Related PTSD (M-PTSD) | 1 year
  The treatment outcome rate was assessed by the Mississippi Scale for Combat-Related PTSD (M-PTSD). A positive outcome rate is represented with the patient post-discharge positive coping, which corresponds to 94-58 points. A treatment failure is regarded as the absent PTSD treatment effect after discharge, which corresponds to 148-113 points and psychic disorders, which correspond to 112-95 points.

CONTACTS AND LOCATIONS:
Overall Officials: Iurii Kuchyn, MD, Study Chair — National medical University named after O. O. Bogomolets, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuchyn IL, Horoshko VR. Predictors of treatment failure among patients with gunshot wounds and post-traumatic stress disorder. BMC Anesthesiol. 2021 Oct 30;21(1):263. doi: 10.1186/s12871-021-01482-8. PMID 34717551